CLINICAL TRIAL: NCT03025711
Title: Use Of Pertuzumab And Trastuzumab Emtansine In Adult Patients With Her2-Positive Metastatic Or Locally Recurrent Unresectable Breast Cancer
Brief Title: Outcomes Of The Spanish Cohort Of Early Access To Pertuzumab And Trastuzumab Emtansine
Acronym: KNOWHER
Status: Completed | Type: Observational
Sponsor: BELEN RUIZ-ANTORAN (Other)
Responsible Party: Sponsor-Investigator, BELEN RUIZ-ANTORAN, Principal Investigator, Puerta de Hierro University Hospital
Organization: Puerta de Hierro University Hospital (Other)
Other Study IDs: ML29844
Record Dates: First submitted 2017-01-11; First posted 2017-01-19 (Estimated); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Breast Neoplasms
Keywords: Advanced HER2+ breast cancer; Pertuzumab; Trastuzumab emtansine; Compassionate use; Early access program; Effectiveness; Safety
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pertuzumab: Patients with HER2-positive metastatic or locally recurrent unresectable breast cancer and who are treated with Pertuzumab under Spanish compassionate use or early access program
- Trastuzumab emtansine: Patients with HER2-positive metastatic or locally recurrent unresectable breast cancer and who are treated with Trastuzumab emtansine (T-DM1) under Spanish compassionate use or early access program

SUMMARY:
The overall study objective is to evaluate the effectiveness and safety of Trastuzumab emtansine (T-DM1) and Pertuzumab under real-world disease conditions in the Spain, and specifically in patients treated under compassionate use or early access program

DETAILED DESCRIPTION:
This is a retrospective, non-interventional, non-comparative, observational cohort study / registry in the Spain. The study design will reflect real-life clinical management of patients with HER2-positive MBC. Type and frequency of actual patient visits and all evaluations will be done as for routine clinical practice.

The analysis of the efficacy and safety results obtained in patients receiving pertuzumab or TDM1 in those early access systems is of utmost importance. These real-world patients with advanced breast cancer may have different characteristics than those enrolled in clinical trials and clinicians must often extrapolate into therapeutic decisions not fully supported by a robust evidence.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18 years at enrolment) with HER2-positive metastatic or locally recurrent unresectable breast cancer and who are treated with Trastuzumab emtansine (T-DM1) or Pertuzumab.
* Patients who initiate Trastuzumab emtansine (T-DM1) and Pertuzumab under Spanish compassionate use or early access program.

Exclusion Criteria:

* Given the characteristics of the study there are no exclusion criteria.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include a cohort of approximately 700 adult patients from the Spain with HER2-positive metastatic or locally recurrent unresectable breast cancer and who are treated with Trastuzumab emtansine (T-DM1) or Pertuzumab under compassionate use or early access program. The decision to initiate use of Trastuzumab emtansine (T-DM1) and Pertuzumab is made independently by the participant and their health care provider and is not mandated by the study design or protocol.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Overall survival. | Through study completion (from date of start of treatment until the date of death from any cause, assessed up to 48 months).
  The time between the date of start of treatment and the date of death. For subjects without documentation of death, OS will be censored on the last date the subject was known to be alive

SECONDARY OUTCOMES:
Progression free survival. | Through study completion (from date of start of treatment until the date of first documented progression assessed up to 48 months)
  The time from start of treatment to the date of the first documented tumour progression as determined by the clinician (may be based on clinical examination or radiographic or laboratory features).
Best overall response rate | Through study completion, an average of 4 year
  Response rate is defined as the proportion of patients with complete response (CR) or partial response (PR) based on their best overall response as written in the medical record
Duration of response (DOR) | Through study completion, an average of 4 year
  The time between the date of first confirmed response to the date of the first documented tumour progression, or death due to any cause, whichever occurs first. At the time of the analysis, several limitations should be taken into consideration for this retrospective study: DOR is only appraisable if measurable disease and DOR data availability in the medical records (ideally assessed with the RECIST criteria) could be incomplete.
Time to treatment failure | Through study completion (from date of start of treatment until the date of treatment failure, assessed up to 48 months)
Time to Objective Response | Through study completion (from date of start of treatment until the date of the first confirmed response, assessed up to 48 months)
  The time from start of treatment to the date of the first confirmed response (evaluated for responders only)
Time to change treatment | Through study completion (from date of start of treatment until the date of change treatment, assessed up to 48 months)
Time to next treatment | Through study completion (from date of start of treatment until the date of start other treatment, assessed up to 48 months)
All suspected Grade 3/4/5 adverse reactions | Through study completion, an average of 4 year
Adverse events of special interest to anti HER2 Mab (AESI) | Through study completion, an average of 4 year
  * AESIs regarding treatment with T-DM1: Hepatic disorder (specific analytical alteration)
  * AESIs regarding treatment with Pertuzumab: Interstitial Lung Disease
AEs of scientific interest | Through study completion, an average of 4 year
  * An asymptomatic decline in LVEF requiring treatment or leading to discontinuation of study treatment (regarding treatment with T-DM1 and Pertuzumab)
  * Other AEs leading to treatment discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Belén Ruiz-Antorán, PhD, Principal Investigator — Department of Clinical Pharmacology, University Hospital Puerta de Hierro Majadahonda, Madrid, Spain
Locations (1):
- Puerta de Hierro University Hospital, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No